CLINICAL TRIAL: NCT00995865
Title: Randomized, Double Blind, Controlled Phase I Trial of the Safety, Tolerability,and Immunogenicity of Graded Doses of XRX-001 Yellow Fever 17D, Inactivated Vaccine, Alum Adsorbed in Healthy Adults.
Brief Title: Trial of Yellow Fever Inactivated Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: X-100-001
Record Dates: First submitted 2009-10-08; First posted 2009-10-15 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Yellow Fever
Keywords: Prevention of yellow fever virus infection
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose (Active Comparator)
  Interventions: Biological: XRX-001 Inactivated yellow fever vaccine
- Mid Dose (Active Comparator)
  Interventions: Biological: XRX-001 Inactivated yellow fever vaccine
- Placebo (Placebo Comparator): NaCl Injectable 0.9%
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: XRX-001 Inactivated yellow fever vaccine — Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL
  Arms: High dose; Mid Dose
Biological: Placebo — NaCl Injectable 0.9%
  Arms: Placebo

SUMMARY:
The Phase 1 trial is a single-center, randomized, double blind, placebo-controlled, dose-ranging out-patient study designed to provide the first clinical data on the safety, tolerability and immunogenicity of XRX-001 inactivated yellow fever vaccine in 60 healthy male and female volunteers, 18-49 years of age. Subjects will receive two inoculations of one of two dose levels of XRX-001 vaccine. A control group will receive placebo.

Safety will be determined by the incidence and severity of adverse events in each treatment group and in the combined cohorts in the double blind treatment period up to 42 days post-vaccination. Subjects will also be followed-up at 3, 6 and 12 months to determine severe adverse events (SAEs) and changes in health status.

Efficacy will be assessed by neutralizing antibody response to the vaccine. The co-primary immunogenicity endpoints will be the dose-response analysis of seroconversion rates (fourfold or greater increase in neutralizing antibody titer between baseline and Day 42) and of the 50% plaque reduction neutralization test (PRNT50) geometric mean titers (GMT) at Day 42.

Secondary immunogenicity endpoints will include:

1. The seroconversion rates and GMT neutralizing antibody titers for all dose groups combined on Days 21 and 42.
2. The reverse cumulative distribution curve of antibody titers on Days 21 and 42 for each dose group and for all dose groups combined
3. The duration of antibody titers displaying the seroconversion rate and GMT across all time-points to Month 12, by treatment group and for both dose groups combined.

ELIGIBILITY:
Inclusion Criteria:

* All aspects of the protocol explained and written informed consent obtained from the subject;
* Aged 18 to 49 years, inclusive;
* In good general health, without significant medical history, physical examination findings, or abnormal laboratory results; and
* Subject must be available for the study duration, including all planned follow-up visits.
* For female subjects of child bearing potential: Negative serum pregnancy tests at Day -7 to -1, and negative urine pregnancy tests prior to vaccination on Days 0, in conjunction with a menstrual and contraceptive history indicating a low probability of pregnancy in the opinion of the physician. Females of childbearing potential will be required to be correctly using an efficacious hormonal method of contraception or intrauterine device for at least 1 month before randomization and during the on-study phase to Day 42. Barrier methods of contraception will not be considered acceptable for study entry. Female subjects of child-bearing potential will acknowledge by signing their informed consent that contraception will be correctly practised during the specified periods and will specify the method used. Female subjects unable to become pregnant must have this documented (e.g. tubal ligation, hysterectomy or postmenopausal [at least one year since last menstrual period]).

Exclusion Criteria:

* History of travel to South America or SubSaharan Africa;
* History of active duty military service;
* History of vaccination against yellow fever, tick-borne encephalitis (TBE), or Japanese encephalitis;
* Went to primary (grade) school in Austria, Germany, Japan, South Korea, India, Thailand, Nepal, Vietnam, or Taiwan (where TBE vaccination is practiced)
* History of dengue fever;
* Known or suspected immunodeficiency disorder, including leukemia, lymphoma, generalized malignancy, or treatment with immunosuppressive medications, including corticosteroids, alkylating agents, antimetabolites, or radiation therapy. Low dose steroids (≤ 10 mg prednisone or equivalent, topical or intra-articular/bursal/tendon/epidural injections of corticosteroids) do not constitute a reason for exclusion;
* History of an autoimmune disorder, including systemic lupus, rheumatoid arthritis, scleroderma, other collagen vascular disease, multiple sclerosis, etc. Psoriasis limited to cutaneous manifestations is not an exclusion criterion;
* Prior history of anaphylaxis to foods, hymenoptera stings, vaccines or drugs;
* Transfusion of blood or treatment with any blood product, including intramuscular or intravenous serum globulin within 3 months of the Screening Visit or anticipated up to Study Day 42;
* Administration of another vaccine within 30 days preceding the screening visit or anticipated up to Day 42 (these subjects may be rescheduled for vaccination at a later date);
* Participation in another clinical trial within 60 days of the screening visit;
* Positive serum or urine pregnancy test prior to vaccination (women of child-bearing potential or lactation or intended pregnancy during study period);
* Abnormalities on laboratory assessment (i.e. meeting the criteria defined for a mild, moderate or severe adverse event in Appendix 1, a1A);
* Seropositive to HIV or HCV or positive for HBsAg;
* Physical examination indicating any clinically significant medical condition;
* Body temperature >38.1°C (100.6°F) or acute illness within 3 days prior to vaccination (subject may be rescheduled);
* Intention to travel out of the area prior to the study visit on Day 42;
* History of excessive alcohol consumption, drug abuse, significant psychiatric illness; and
* Intention to increase normal exercise routine, participate in contact sports or strenuous weight lifting or to initiate vigorous exercise from Screening until after Day 42.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanada Culliton, Study Director — GE Healthcare Bio-Sciences
Locations (1):
- Johnson County Clin-Trials, Lenexa, Kansas, United States

REFERENCES:
- [Derived] Monath TP, Fowler E, Johnson CT, Balser J, Morin MJ, Sisti M, Trent DW. An inactivated cell-culture vaccine against yellow fever. N Engl J Med. 2011 Apr 7;364(14):1326-33. doi: 10.1056/NEJMoa1009303. PMID 21470010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 of the Subjects in the High-Dose made it thru the study, however, it was later found that those 2 subjects vaccinated prior to joining this study. One (1) subject in the "Placebo" went thru the the study, but was later lost to follow-up.
Pre-assignment Details: 60 Subjects enrolled in this study. 3 Subjects discontinued in this study.
Period: Overall Study
Arm/Group | High Dose | Mid Dose | Placebo
Started | 24 | 24 | 12
Completed | 22 | 24 | 11
Not Completed | 2 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Dose Group: Two groups of 24 subjects each, (one arm called a high dose group, the other a Mid-Dose group) were to receive two intramuscular (IM) injections (0.5mL) of XRX-001 vaccine containing either greater than or equal to 8.0 log10 VE/dose (viral equivalent) (high dose) or 1/10th of the high dose for the (mid dose).
- Mid-Dose Group: Two groups of 24 subjects each were to receive two intramuscular (IM) injections (0.5mL) of XRX-001 vaccine containing either greater than or equal to 8.0 log10 VE/dose (viral equivalent) (high dose) or 1/10th of the high dose for this (mid dose) group.
- Placebo Group: This third group of 12 subjects were to receive a placebo (0.9% normal saline for injection).
- Total: Total of all reporting groups
Arm/Group | High Dose Group | Mid-Dose Group | Placebo Group | Total
Number analyzed (Participants) | 22 | 24 | 11 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 11 | 57
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.0) | 31 (9.1) | 29 (8.2) | 32 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 6 | 25
  Male | 13 | 14 | 5 | 32
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 11 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Incidence and Severity of Adverse Events in Each Treatment Group in the Double-blind Treatment Period up to 42 Days Post-vaccination.
Description: Subjects were observed for 60 minutes (greater than of equal to 60 minutes and less than of equal to 90 minutes) after vaccine adminstration for any signs or symptoms or local and/or systematic intolerance to the test articles and vital signs were to be checked within the same observation timeframe.
  After vaccination, subjects were to complete a memory aid to record daily temperature, symptoms, and concomitant medications from Day-0 to Day-42.
  Subjects were to return to the clinic on Days 3, 10, 21, 24, 31, and 42 with a second vaccination given on Day 21.
  At each visit, study personnel were to conduct a structured adverse event (AE) interview, and subject were to use their memory aid to assist with the recall of symptoms experiences and daily oral temperatures.
Time Frame: Measured from 0 up to 21 Days
Population: Subjects were to return to the clinic on Days 3,10, 21, 24, 31,and 42 with the second vaccination given on Day 21. At each visit, study personnel were to conduct a structured adverse event (AE) interview, and subject were to use their memory aid to assist with the recall of symptoms experiences and daily oral temperatures.
Measure: Number; unit: participants
Groups:
- High Dose Group: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL.
  24 Subjects were examined in this group.
- Mid Dose Group: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL
- Placebo Group: Subjects were administered with NaCl Injectable 0.9%.
  12 Subjects were examined in this group.
Arm/Group | High Dose Group | Mid Dose Group | Placebo Group
Number analyzed (Participants) | 24 | 24 | 12
participants
  Days 0-21 (1st injection)-Pain | 13 | 13 | 2
  Days 0-21 (1st injection)-Redness | 22 | 21 | 10
  Days 0-21 (1st injection)-Tenderness | 15 | 19 | 4
  Days 0-21 (1st injection)-Swelling | 22 | 21 | 10
  Days 0-21 (1st injection)-Itching | 3 | 1 | 0
  Days 0-21 (1st injection)-Diarrhea | 0 | 4 | 3
  Days 0-21 (1st injection)-Malaise | 4 | 2 | 3
  Days 0-21 (1st injection)-Headache | 2 | 8 | 7
  Days 0-21 (1st injection)-Tiredness | 7 | 2 | 5
  Days 0-21 (1st injection)-Nausea | 3 | 0 | 1

2. Secondary Outcome: Percentage of Subjects With Seroconversions or Who Are Seropositive Using 2 Dose Levels of XRX-001
Description: Secondary immunogenicity endpoints will use 2 dose levels of XRX-001 inactivated yellow fever vaccine determined by 50% plaque reduction neutralization test (PRNT50). Dose groups were to be compared for neutralizing antibody seroconverison rate, distribution of antibody titers, and geometric mean antibody titers (GMTs) to yellow fever 17D virus. The seroconversion rates and GMT neutralizing antibody titers for each dose group and all dose groups combined; The reverse cumulative distribution curve of antibody titers;
Time Frame: Days 21 and 42, 12 months
Population: Seropositive was to show a significant level of serum antibodies, or other immunologic marker in the serum, indicating previous exposure to the infectious agent being tested. In immunology, seroconversion is the time period during which a specific antibody develops and becomes detectable in the blood.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- High Dose Group; Mid Dose Group: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL
- Placebo Group: NaCl Injectable 0.9%
  Placebo: NaCl Injectable 0.9%
Arm/Group | High Dose Group | Mid Dose Group | Placebo Group
Number analyzed (Participants) | 22 | 24 | 11
Percentage of subjects
  Seropositive-Day 21(21 Days after 1st Injection) | 46 [24 to 68] | 13 [3 to 32] | 0 [0 to 29]
  Serocovert-Day 21 (21 Days after 1st Injection) | 32 [14 to 55] | 13 [3 to 32] | 0 [0 to 29]
  Seropositivity-Day 31 (10 Days after second Inj) | 100 [85 to 100] | 88 [68 to 97] | 0 [0 to 29]
  Seroconvert- Day 31 (10 Days after second Inj) | 100 [85 to 100] | 75 [53 to 90] | 0 [0 to 29]
  Seropositivity -Day 42 (21 Days after 2nd Inj) | 100 [85 to 100] | 88 [68 to 97] | 0 [0 to 29]
  Seroconvert-Day 42 (21 Days after 2nd Inj) | 100 [85 to 100] | 71 [49 to 87] | 0 [0 to 29]

3. Secondary Outcome: Distribution of Geometric Mean Antibody Titers (GMTs) to Yellow Fever 17D Virus.
Description: Geometric mean antibody titers (GMT) neutralizing antibody titers for each dose groups.
Time Frame: GMT titers measured at days 21, 31 and 42 for different dose rates.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Antibody titers
Arm/Group | High Dose Group | Mid Dose Group | Placebo Group
Number analyzed (Participants) | 22 | 24 | 11
Geometric Antibody titers
  Geometric mean titer Day 21--21 Days 1st Inj) | 10 [7 to 15] | 6 [5 to 8] | 5 [5 to 5]
  Geometric mean titer Day 31--10 Days after 2nd Inj | 146 [104 to 203] | 39 [22 to 69] | 5 [5 to 5]
  Geometric mean titer Day 42--21 Days after 2nd Inj | 113 [81 to 159] | 30 [18 to 49] | 5 [5 to 5]

4. Primary Outcome: The Incidence and Severity of Adverse Events in Each Treatment Group in the Double-blind Treatment Period up to 42 Days Post-vaccination.
Description: as for outcome 1
Time Frame: Measured from 22 up to 42 Days.
Population: Subjects were to combined at days 22 to 42 . At each visit, study personnel were to conduct a structured adverse event (AE) interview, and subject were to use their memory aid to assist with the recall of symptoms experiences and daily oral temperatures.
Measure: Number; unit: participants
Arm/Group | High Dose Group | Mid Dose Group | Placebo Group
Number analyzed (Participants) | 24 | 24 | 12
participants
  Days 22-42 (2nd injection)-Pain | 6 | 8 | 0
  Days 22-42 (2nd injection)-Tenderness | 8 | 10 | 0
  Days 22-42 (2nd injection)-Redness | 12 | 16 | 7
  Days 22-42 (2nd injection)-Swelling | 12 | 16 | 7
  Days 22-42 (2nd injection)-Vomiting | 1 | 2 | 3
  Days 22-42 (2nd injection)-Malaise | 1 | 4 | 5
  Days 22-42 (2nd injection)-Headache | 1 | 6 | 5
  Days 22-42 (2nd injection)-Muscle Ache | 0 | 3 | 3
  Days 22-42 (2nd injection)-Feverishness | 0 | 3 | 3
  Days 22-42 (2nd injection)-Chills | 0 | 2 | 1
  Days 22-42 (2nd injection)-Tiredness | 2 | 4 | 4
  Days 22-42 (2nd injection)-Nausea | 1 | 3 | 3
  Days 22-42 (2nd injection)-Drowsiness | 1 | 5 | 3
  Days 22-42 (2nd injection)-Shortness of Breath | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Two intramuscular injections at an interval of 21 days
Description: Two intramuscular injections at an interval of 21 days. First injection administered on day with an interval of 21 days followed by a second injection on day 22.
Groups:
- High Dose First Injection; Mid Dose First Injection: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL.
  First injection.
- Placebo First Injection: NaCl Injectable 0.9%
  Placebo: NaCl Injectable 0.9% First injection.
- High Dose Second Injection: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL.
  Second injection at an interval of 21 days
- Mid Dose Second Injection: XRX-001 Inactivated yellow fever vaccine: Inactivated yellow fever vaccine, alum adsorbed, High dose = 2.3 x 10^8 VE/0.5mL and Mid dose = 2.2 x 10^7 VE/0.5mL.
  Second injection.
- Placebo Second Injection: NaCl Injectable 0.9%
  Placebo: NaCl Injectable 0.9% Second injection.
Arm/Group | High Dose First Injection | Mid Dose First Injection | Placebo First Injection | High Dose Second Injection | Mid Dose Second Injection | Placebo Second Injection
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/12 | 0/24 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 24/24 | 24/24 | 12/12 | 24/24 | 24/24 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose First Injection (N=24) | Mid Dose First Injection (N=24) | Placebo First Injection (N=12) | High Dose Second Injection (N=24) | Mid Dose Second Injection (N=24) | Placebo Second Injection (N=12)
Pain at Injection site (Skin and subcutaneous tissue disorders) | 13 (13) | 13 (13) | 2 (2) | 6 (6) | 8 (8) | 0 (0) — General pain at the site of injection
Tenderness at injection site (Skin and subcutaneous tissue disorders) | 15 (15) | 19 (19) | 4 (4) | 8 (8) | 10 (10) | 0 (0) — Tenderness at the site of injection
Redness at Site of Inection (Skin and subcutaneous tissue disorders) | 22 (22) | 21 (21) | 10 (10) | 12 (12) | 16 (16) | 7 (7) — Redness at the site of injection
Swelling at site of injection (Skin and subcutaneous tissue disorders) | 22 (22) | 21 (21) | 10 (10) | 12 (12) | 16 (16) | 7 (7) — Swelling at the site of injection
Itching at site of ijnection (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Itching a the site of injection
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Diarrhea
Malaise (General disorders) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 5 (5) — Malaise
Headache (General disorders) | 2 (2) | 8 (8) | 7 (7) | 1 (1) | 6 (6) | 5 (5) — Headache
Tiredness (General disorders) | 7 (7) | 2 (2) | 5 (5) | 2 (2) | 4 (4) | 4 (4) — Tiredness
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) — Nausea
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) — Vomiting
Muscle Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) — Muscle Ache
Feverishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) — Feverishness
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Chills
Drowsiness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) — Drowsiness
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Shortness of Breath

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No